CLINICAL TRIAL: NCT05635500
Title: Clinical Comparison Between Midline and Right-sided Insertion of the Videolaryngoscope for Intubation - a Randomized, Controlled, Prospective Clinical Trial
Brief Title: Clinical Comparison Between Midline and Right-sided Insertion of the Videolaryngoscope for Endotracheal Intubation
Acronym: Midway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sascha Treskatsch, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EA2/121/21
Record Dates: First submitted 2021-07-22; First posted 2022-12-02 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Intervention Model Description: Computer generates randomisation in two groups middle insertion (n=92) and right insertion (n=92)
Who Masked: Participant
Masking Description: Computer generated randomisation, Patient under general anaesthesia during procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Middle Insertion (Experimental): Videolaryngoscope is inserted from the middle for endotracheal intubation.
  Interventions: Procedure: Different Approach to endotracheal intubation.
- Right Insertion (No Intervention): Videolaryngoscope is inserted from the right for endotracheal intubation.

INTERVENTIONS:
Procedure: Different Approach to endotracheal intubation. — Different insertion way.
  Arms: Middle Insertion

SUMMARY:
The videolaryngoscope is an established tool for securing the airway, even in difficult situations. It remains unclear which insertion technique is the safest and fastest in the difficult airway.

DETAILED DESCRIPTION:
Videolaryngoscopy is one of the standard methods of airway management in the Department of Anesthesiology with Surgical Intensive Care, is anchored in the applicable Standard Operating Procedures (SOP) and is used in everyday clinical practice.

In order to establish the above-mentioned generality, the patients are divided into 2 groups. In the preoperative visit, the patients are divided into easy and difficult airway, and a randomization regarding the induction technique is done paper-based after induction of anesthesia.

Patients* identified in the preoperative visit with a risk for difficult intubation or difficult laryngoscopy (Mallampati ≥ 3, thyromental distance below 6.5cm, sternomental distance below 12.5cm, conversion from conventional laryngoscopy to VLS in the history, cervical spine immobilization, lack of possibility for reclination) are randomized into one of the two groups:

Group DR (difficult right) corresponds here to the right-sided insertion technique in the difficult airway.

Group DM (difficult middle) corresponds to the middle access route in the difficult airway.

Perioperatively, standard monitoring is performed according to the hospital's SOP, consisting of a 3-point ECG recording, non-invasive blood pressure measurement, pulse oximetry, respiratory gas monitoring and the recording of a processed EEG for hyponosis depth measurement. To ensure and document optimal muscle relaxation, we perform relaxometry.

In accordance with the hospital's internal SOP, anesthesia induction is performed after sufficient preoxygenation with opiates, hypnotics and muscle relaxants. All drugs are administered in accordance with the operation-specific, internal hospital standards.

In addition to the basic measures, the standardized, extended measures for the management of a difficult airway are all fulfilled in the DR and DM groups and documented by means of a checklist. These include optimized positioning and adequate depth of anesthesia, as well as the provision and use of various aids such as a guide rod or frovacatheter.

Prior to videolaryngoscopy, a mouth guard is inserted unless contraindicated for airway protection.

This is followed by videolaryngoscopy with insertion of the videolaryngoscope according to the assigned group, and then insertion of the endotracheal tube.

The visualization of the laryngeal plane using the Cormack/Lehane score, Video Classification of Intubation (VCI) score and the different process times of airway protection are documented in addition to the vital signs and train-of-four (TOF).

In addition to the video laryngoscope to optimize visualization, standardized advanced techniques for laryngoscopy as well as for intubation are used and documented if necessary.

In addition, the anatomic, pathologic, and other typical conditions that caused the current difficult intubation are documented.

The laryngoscopy including intubation is recorded via the VLS in the form of a video. This allows an assessment of the visual scores by an independent observer*. Blinding cannot take place due to the different insertion techniques. The video recording only shows the inside of the mouth and larynx.

Side effects/complications are recorded on the 1st postoperative day by means of a short visit and standardized questionnaire according to localization (sore throat, hoarseness, mucosal lesions, dysphagia, dental damage) and differentiated according to the extent to which these complaints can be attributed to the surgical intervention and/or airway protection.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery under general anesthesia with indication for airway protection via endotracheal intubation
* age ≥ 18 years
* indication for primary videolaryngoscopic Intubation (VLS) and/or at least one of the following criteria:

  1. Mallampati ≥ 3
  2. Thyromental distance <6.5cm
  3. Sternalomental distance <12.5 cm
  4. Conversion from conventional laryngoscopy to VLS in history
  5. Cervical spine immobilization/lack of ability to recline.

Exclusion Criteria:

* Pregnant patients
* Participation in another prospective clinical intervention study within the last 30 days and during participation in this study
* Necessary Rapid Sequence Induction
* Indications of impossible mask ventilation and/or videolaryngoscopy (mouth opening < 3.5 cm, ...)
* Existence of tracheal cannula prior to operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Comack-Lehane Classification | immediately after the intervention
  Laryngeal vision is determined by Cormack/Lehane classification (C/L)

SECONDARY OUTCOMES:
Time to intubate | immediately after the intervention
  Defined as time between endotracheal tube passing the lips till blocking of the cuff.
First pass success | immediately after the intervention
  Defined as no further attempts has been taken.
Time to laryngeal view | immediately after the intervention
  Defined as time from the insertion of the laryngoscope till position of the best overview of the larynx.
Complications during induction | 15 minutes
  Defined as hemodynamic changes (bradycardia < 60 bpm, tachycardia >100 bpm, hypotension < 65 mmHG MAD, hypertension > 100 mmHG MAD), Oxygendesaturation <92 % SpO2, the need for further equipment (e.g. flexible bronchoscope), bleedings or a surgical airway
Complication on first postoperative day | 24 hours
  Definde as the occurence of swelling, bleedings, damage on teeth, throat hoarseness

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Department of Anesthesia and operative intensive Care, Campus Benjamin Franklin, Charité - University Hospital Berlin, Steglitz, State of Berlin
  - Campus Benjamin Franklin, Charité - Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang L, Qiu S, Zhang P, Yao W, Chang Y, Dai Z. The midline approach for endotracheal intubation using GlideScope video laryngoscopy could provide better glottis exposure in adults: a randomized controlled trial. BMC Anesthesiol. 2019 Nov 5;19(1):200. doi: 10.1186/s12871-019-0876-6. PMID 31690285